CLINICAL TRIAL: NCT05915754
Title: Effects of Posterior Oblique Sling Strengthening Exercises on Pain & Flexibility Among Runners With Iliotibial Band Syndrome
Brief Title: Effects of Posterior Oblique Sling Strengthening Exercises on Pain & Flexibility Among Runners With
Acronym: ITBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REC/RCR&AHS/23/0420
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Iliotibial Band Syndrome
Keywords: lateral knee pain, Posterior Oblique Sling, Runner
MeSH Terms: conditions — Iliotibial Band Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip abductors stretching and strengthening exercises (Experimental): Patients will get the hip abductor stretching and strengthening exercise treatment for four weeks four times per week and will consist of four sets of 15 repetitions.
  Interventions: Other: Hip abductors stretching and strengthening exercises
- Posterior oblique sling strengthening exercises (Experimental): Patients will get treatment plan of Hip abductors stretching and strengthening exercises plus a posterior oblique sling strengthening program for four weeks, four times per week and will consist of four sets of 15 repetitions.
  Interventions: Other: Posterior oblique sling strengthening exercises

INTERVENTIONS:
Other: Hip abductors stretching and strengthening exercises — Treatment consist of four stretches for the ITB including: ITB stretch with trunk side bend, ITB stretch with trunk side bend and upward lateral reach, trunk side bend with downward lateral reach and side lying leg adduction and Strengthening exercise plan involving the gluteal muscle groups. These exercises include clams, side-lying abduction, reverse clams and supine bridge
  Arms: Hip abductors stretching and strengthening exercises
Other: Posterior oblique sling strengthening exercises — Treatment consists of treatment A plus the intervention program of POSS consisted of four different exercises utilizing activation of the POSS. The intervention program focuses on one specific exercise each week that will progress in difficulty over the 4 weeks. The equipment used in the exercise progression included a blue, latex-free, medium-resistance theraband (TB), and the final exercise of the progression will include the use of a step stool. The TB will be used to increase the activation of the latissimus dorsi while simultaneously performing lower-extremity exercise to increase gluteal muscle involvement. The exercises are to be used in the 4-week progression.
  Arms: Posterior oblique sling strengthening exercises

SUMMARY:
The popularity of recreational running and rate of running related injuries are increasing. Research has shown that iliotibial band syndrome (ITBS) is one of the most common knee injuries among runners alongside plantar fasciitis, meniscal injuries, patellar tendinopathy, and patelleofemoral pain (PFP). ITBS is twice as common in female runners as compared to male long distance runners due to biomechanical variations. Literature supports the use of gluteal strengthening and IT band stretching as an effective treatment for iliotibial band syndrome. Posterior oblique sling is activated during running and its weakness is thought to be the predisposing factor of iliotibial band syndrome among long distance runners. The purpose of this study is to evaluate the effectiveness of posterior oblique sling exercises in decreasing lateral knee pain and improving flexibility of iliotibial band among female runner compared to gluteal strengthening and IT band stretching alone.

Data will be collected by using non-probability purposive sampling method. Sample size will be 26. 13 Female runners with average running of 15 kilometers per week and chronic iliotibial band syndrome will be employed in two different study groups A and B randomly. Both groups will get treatment for four weeks four times per week. Control group A will get conventional treatment of hip abductors strengthening and Iliotibial band stretching and Experimental group B will get posterior oblique sling strengthening exercises plus conventional hip abductors strengthening and IT band stretching. Pain and flexibility will be measured before treatment after every week and by the end of the month to note progression. Numeric Pain Rating Scale (NPRS) will be used to rate pain and modified Ober's test using digital inclinometer will be used to rate flexibility of iliotibial band. Statistical analysis will be done using SPSS latest version

DETAILED DESCRIPTION:
The purpose of this study is to compare the two different treatment protocols for Iliotibial band syndrome and help create an effective treatment option for long distance runners who suffer lateral knee pain due to IT band tightness.

The study will be Randomized control trial. Non-probability purposive sampling method will be used.Subjective and objective data of all the participants will be taken by using NPRS, Modified Ober's test using Digital inclinometer, Noble's compression test and ITB Questionnaire.

Researcher will take careful history of the participant with proper assessment and examination of the knee.

At baseline, weekly and by the end of 4th week of treatment objective and subjective measurements of participants will be taken using NPRS, Modified Ober's test using Digital inclinometer, Noble's Compression test and ITB Questionnaire.

All the participants will receive equal treatment of 4 weeks. The Data will be analyzed using SPSS for windows software version 25. Statistical significance P=0.05. After assessing the normality of current data by shapiro wilk test. it will be decided whether parametric or non parametric test will be used within the groups or between 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Female Treadmill runners of age 18 to 35 years.
* Perform running of average 15 running kilometers per week and Experience of burning lateral knee pain after 2nd-3rd kilometer of running
* Localized point tenderness over the femoral condyle about 2-4 cm above joint line on palpation
* Positive Noble's Compression test
* Positive modified Ober's Test

Exclusion Criteria:

* Short distance runners
* People with any other medical condition Including myofacial pain syndrome, early degenerative joint disease, lateral collateral ligament pathology, lateral meniscal injuries, tibiofibular joint sprain, popliteal or biceps femoris tendonitis, or referred pain from lumbar spine. All these conditions will be ruled out with carefully history and examination
* People taking any other form of treatment including corticosteroids, non-steroidal anti-inflammatory drugs or analgesics
* People with previous history of surgical treatment for ITBS
* People with neurological deficits or systemic illness

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-06-25 (Estimated); Study Completion 2023-07-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale-101 Questionnaire: | 4 weeks
  The patient's perception of their pain intensity level is recorded on a numerical scale from 1 to 100, with 0 being no pain and 100 being the worst pain. The patient indicates by means of a percentage on a 10cm line, when the pain was at its worst and again on another 10cm line when the pain was at its least. The average of these two figures indicates the average pain experienced by the patient as a percentage. NRS-101 questionnaire is regarded as a superior measuring instrument, being extremely easy to administer and score. It can be done either in written or verbal form, or due to its simplicity, there are very low tendencies for incorrect responses from patients.
Modified Ober's test using digital inclinometer | 4 weeks
  ITB tightness is elicited by this test and will be measured using digital inclinometer.The use of an inclinometer to measure hip adduction using both the Ober test and the modified Ober test appears to be a reliable method for the measurement of ITB flexibility. As described the test is performed as follows: The patient is made to lie laterally recumbent with the affected side uppermost. The affected lower limb was then brought into full extension by the examiner, with some abduction at the hip. In the Ober's test, the knee is flexed at this moment during the test, while in the Modified Ober's test, the knee is left extended. The examiner then slowly releases support of the limb, allowing the limb to fall into adduction past the neutral position. This constitutes a normal or negative test. A tight ITB restricts adduction and prevents the knee from falling past the neutral position. This constitutes a positive test for ITB tightness
Noble's Compression test: | 4 weeks
  The test is performed as follows: The patient is made to lie supine with the affected knee flexed to 90 degrees. Pressure is placed over the proximal part of the lateral femoral condyle. The knee was then gradually extended, and at 30 to 40 degrees, if the patient complained of a similar pain to that experienced while running, then the test was positive for ITBS
ITB Questionnaire | 4 weeks
  The effect on participants' running performance will be measured using the ITB Questionnaire. The ITB Questionnaire was designed by the author of the study (Wood, 1997) for the measurement of patient disability specifically for ITBS.
The Daily Exercise Diary | 4 weeks
  The Daily Exercise Diary will be used to monitor participant compliance and ability to perform the exercises. The Daily Exercise Diary was designed by the author of the study (Wood, 1997) for the measurement of patient disability specifically for ITBS.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Nosheen Manzoor, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- SHAPES gymnasium, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foch E, Reinbolt JA, Zhang S, Fitzhugh EC, Milner CE. Associations between iliotibial band injury status and running biomechanics in women. Gait Posture. 2015 Feb;41(2):706-10. doi: 10.1016/j.gaitpost.2015.01.031. Epub 2015 Feb 7. PMID 25701012
- [Background] Charles D, Rodgers C. A LITERATURE REVIEW AND CLINICAL COMMENTARY ON THE DEVELOPMENT OF ILIOTIBIAL BAND SYNDROME IN RUNNERS. Int J Sports Phys Ther. 2020 May;15(3):460-470. PMID 32566382
- [Background] Gordon S. Iliotibial Band Syndrome. Clinical Practice Guidelines. 2018:321.
- [Background] Fredericson M, Wolf C. Iliotibial band syndrome in runners: innovations in treatment. Sports Med. 2005;35(5):451-9. doi: 10.2165/00007256-200535050-00006. PMID 15896092
- [Background] van der Worp MP, van der Horst N, de Wijer A, Backx FJ, Nijhuis-van der Sanden MW. Iliotibial band syndrome in runners: a systematic review. Sports Med. 2012 Nov 1;42(11):969-92. doi: 10.2165/11635400-000000000-00000. PMID 22994651
- [Background] Mouw J. The Effects of Posterior Oblique Sling Exercises on a Runner with Iliotibial Band Syndrome: Azusa Pacific University; 2019.
- [Background] McKay J, Maffulli N, Aicale R, Taunton J. Iliotibial band syndrome rehabilitation in female runners: a pilot randomized study. J Orthop Surg Res. 2020 May 24;15(1):188. doi: 10.1186/s13018-020-01713-7. PMID 32448384
- [Background] Gangat AK. The effectiveness of gluteus medius and iliotibial band stretching, versus strengthening, in the rehabilitation of iliotibial band syndrome in long distance runners. 2005.
- [Background] Baker RL, Fredericson M. Iliotibial Band Syndrome in Runners: Biomechanical Implications and Exercise Interventions. Phys Med Rehabil Clin N Am. 2016 Feb;27(1):53-77. doi: 10.1016/j.pmr.2015.08.001. PMID 26616177
- [Background] SieunNarine-McKay J. Evaluation of outcomes in assessment of iliotibial band syndrome rehabilitation programs: University of British Columbia; 2016
- [Background] Rosenthal MD. Clinical testing for extra-articular lateral knee pain. A modification and combination of traditional tests. N Am J Sports Phys Ther. 2008 May;3(2):107-9. PMID 21509133
- [Background] Kahl C, Cleland JA. Visual analogue scale, numeric pain rating scale and the McGill Pain Questionnaire: an overview of psychometric properties. Physical therapy reviews. 2005;10(2):123-8.
- [Background] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962
- [Background] Kesminas R, Burbulevičiūtė J. Ober's Test and Modified Ober's Test are Reliable Means of Measuring Iliotibial Band using both Goniometer and Inclinometer. Reabilitacijos mokslai: slauga, kineziterapija, ergoterapija. 2019;2
- [Background] Colaco J, Dudley N, Karmacharya N, Holbein-Jenny M. Interrater reliability and validity of Ober's, Noble compression, and modified Thomas tests. Physical therapy. 2002:5-8